CLINICAL TRIAL: NCT01435681
Title: Can Short Latency Afferent Inhibition Give us Clues to Better Dystonia Treatments?
Brief Title: Can Short Latency Afferent Inhibition Give us Clues to Better DYT 1 Dystonia Treatments?
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Brain and Spinal Cord Injury Research Trust Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 405-2011
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: DYT-1; DYT1; DYT 1; Dystonia
Keywords: DYT-1; DYT1; DYT 1; dystonia; DBS; deep brain stimulation; TMS; transcranial magnetic stimulation
MeSH Terms: conditions — Dystonia musculorum deformans type 1; Dystonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DYT-1 Postive: This group includes those participants who enroll having a genetically confirmed primary generalized dystonia diagnosis.
- Control: This group includes healthy subjects between the ages of 18 and 80.

SUMMARY:
This is a research study using transcranial magnetic stimulation (TMS) to investigate interactions between the sensory system and the motor cortex in primary generalized dystonia (DYT1 dystonia) subjects who undergo deep brain stimulation (DBS) surgery.

The sensory system is the body's sense organs - smell, sight, sound, etc. - and the motor cortex is the part of your brain where nerve impulses control voluntary muscle activity.

DETAILED DESCRIPTION:
The cause of DYT1 dystonia is not clear. DYT1 dystonia symptoms include abnormal posture or repetitive twisting movements affecting one body part; in some patients, the entire body can twist and contort painfully. Magnetic resonance imaging (MRI) studies are normally used to evaluate changes in brain structure in DYT1 dystonia. Transcranial magnetic stimulation (TMS) is a painless, non-invasive method to test how your brain conducts electrical messages to the rest of your body, including your muscles.

If you are a DYT1 dystonia patient, then this study involves up to three visits. The first visit (before DBS surgery) will last about 4 hours and the second and third visits (after DBS surgery) will last about 4 hours as well. These visits will include a complete physical and neurological exam, video recorded dystonia and mood rating scales, followed by electromyography (EMG) and TMS sessions. Subjects who have already undergone DBS surgery may participate in applicable visits based on the length of time since their DBS surgery.

If you are a control subject, this study involves one visit, about 4 hours long. This visit will include TMS and EMG sessions.

ELIGIBILITY:
INCLUSION CRITERIA:

* Between the ages of 10 and 80 years. (CONTROL SUBJECTS between 18-80 years)
* Diagnosis and genetic test results confirming diagnosis of DYT1 dystonia.
* Currently treated with medications and enrolled in evaluation process for DBS surgery to confirm candidacy - OR -
* Previous DBS surgery

EXCLUSION CRITERIA:

* Implanted pacemaker, medication pump, vagal stimulator, Transcutaneous electrical nerve stimulation (TENS) unit or ventriculoperitoneal shunt.
* Family or personal history of medication refractory epilepsy.
* Pregnancy: due to the frequent visits over a prolonged period and the lack of Information on the safety of TMS during pregnancy, pregnant women will not be eligible to participate in this study. Women of childbearing potential will be eligible to participate, provided that they are using adequate contraception during TMS treatments.

This study is accepting healthy volunteers, aged 18-80, as control subjects. Control subjects will not undergo DBS surgery.

EXCLUSION CRITERIA (as it applies to healthy control subjects):

* Cannot have family history or personal history of medication refractory epilepsy

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects scheduled to undergo pallidal deep brain stimulation surgery for DYT1 dystonia will be enrolled up to 12 months for this pilot trial. Genetic test results confirming DYT1 gene mutation will be reviewed prior to consenting research subjects. Patients who are diagnosed with DYT1 dystonia and are candidates for DBS surgery will be indentified as candidates for the research study. Additionally, subjects who have already undergone DBS surgery will be identified as candidates.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in amplitude, at 3 and 6+ months, of motor evoked potentials (MEPs) with median nerve stimulation (SAI) and simultaneous median nerve and ulnar nerve stimulation (SAIdualstim) | 3 and 6+ months post-DBS surgery
  Surface electromyography (EMG) will be recorded from the first dorsal interosseous muscle to determine the amplitude of potentials evoked in two ways - SAI and SAIdualstim. For SAI, potentials will be evoked with median nerve stimulation preceding TMS by the N20 latency plus 3 ms. For SAI dualstim, simultaneous stimulation of median and ulnar nerves will precede TMS by the N20 latency plus 3 ms.

SECONDARY OUTCOMES:
Correlation of change in evoked potential amplitudes and clinical measures at 3 and 6+ months | 3- and 6+-months post-DBS surgery
  The changes, from baseline to 3 and 6+ months post-operation, in amplitudes recorded during SAI and SAIdualstim testing will will be correlated with the changes in the clinical measures taken at the same timepoints. The Spearman correlation test will be used for this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle Shukla, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: UF Center for Movement Disorders & Neurorestoration — http://movementdisorders.ufhealth.org/